CLINICAL TRIAL: NCT03812003
Title: Investigation of the Strategy of Preventing Post-operative Opioid-induced Hyperalgesia by Remifentanil Infusion
Brief Title: Investigation of the Strategy of Preventing Post-operative Opioid-induced Hyperalgesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hung Chan, Principal Investigator, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2-107-05-162
Record Dates: First submitted 2019-01-13; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Opioid-Induced Disorders
Keywords: opioid-induced hyperalgesia, remifentanil
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Intervention Model Description: Breast cancer patient
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- remifentanil (Experimental): After emergence and extubation of endotracheal tube, remifentanil 1mcg/kg were diluted with 0.9% saline to 50 ml, added in IV bag, and drip for 30 minutes.
  Interventions: Drug: Remifentanil
- no intervention (No Intervention): After emergence and extubation of endotracheal tube, 0.9% saline 50ml were added in IV bag and drip for 30 minutes.

INTERVENTIONS:
Drug: Remifentanil — remifentanil 1mcg/kg added in 0.9% saline and diluted to 50ml
  Other Names: Remifentanil ALVOGEN powder
  Arms: remifentanil

SUMMARY:
The concept of Enhanced Recovery After Surgery(ERAS) has been prevalent in recent years. In the ERAS guideline, short-acting anesthetics, instead of long-acting opioid anesthetics, were recommended during surgery to decrease post-operative complication and length of hospital stay. Propofol-remifentanil based total intravenous anesthesia (TIVA) can provide quicker emergence and decreased post-operative nausea and vomiting. However, the prescription of opioid (especially remifentanil) may induce opioid-induced hyperalgesia (OIH) and increase the requirement of analgesics. Previous studies provided some strategies to prevent OIH. The purpose of this study is to investigate the effect of adding remifentanil(1 mcg/kg) after emergence and endotracheal extubation in breast cancer females receiving breast surgery under propofol-remifentanil based TIVA for the prevention of OIH.

DETAILED DESCRIPTION:
1. After obtaining informed consent, patients will be randomized into two groups.
2. All patients receive remifentanil-propofol based TIVA and Bispectral index (BIS) monitor during breast surgery. In the end of surgery, intravenous NSAID(keto) 30mg and local anestehsia (Marcaine) infiltration around the surgical wound will be prescribed to reduce post-operative pain.
3. group R(intervention): remifentanil 1mcg/kg diluted with 0.9% saline to 50ml and drip for 30 minutes after emergence and extubation of endotracheal tube
4. group N(no intervention): 0.9% saline 50ml drip for 30 minutes after emergence and extubation of endotracheal tube
5. In post-anesthesia room: record the numerical rating scale (NRS); requirement of additional analgesics (rescue medication), blood pressure, heart rate, pulse oximeter, degree of nausea, vomiting
6. In ward: record the numerical rating scale (NRS) and total analgesics consumption

ELIGIBILITY:
Inclusion Criteria:

* Subject's ASA (American Society of Anesthesiologists) Physical Status Classification: I (A normal healthy patient)~III(A patient with severe systemic disease)
* Subject has breast cancer and scheduled for breast surgery using total-intravenous anesthesia(TIVA)

Exclusion Criteria:

* Subject's ASA (American Society of Anesthesiologists) Physical Status Classification >3
* Subject doesn't receive total-intravenous anesthesia(TIVA) during surgery
* Subject has psychiatric disease
* allergic to opioid or propofol
* History of alcoholism
* History of drug abuse

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — breast cancer female
Enrollment: 100 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Score (NRS) for pain score in post-anesthesia room (PAR) | 0 minutes
  1.The pain after breast surgery is moderate and suppose to be reduced after combined prescription of NSAID and local analgesics. Post-operative pain is supposed to be related with hyperalgesia. 2.Record the degree of post-operative pain by Numerical Rating Scale (Numerical Rating Scale)(0-10; 0= no pain; 10=pain as bad as can be)
Numerical Rating Score (NRS) for pain score in post-anesthesia room (PAR) | 30 minutes
  1.The pain after breast surgery is moderate and suppose to be reduced after combined prescription of NSAID and local analgesics. Post-operative pain is supposed to be related with hyperalgesia. 2.Record the degree of post-operative pain by Numerical Rating Scale (Numerical Rating Scale)(0-10; 0= no pain; 10=pain as bad as can be)
The amount analgesic requirement in post-anesthesia room (PAR) | 30 minutes
  1.The pain after breast surgery is moderate and suppose to be reduced after combined prescription of NSAID and local analgesics during surgery. Post-operative pain is supposed to be related with hyperalgesia. 2.Record the degree of post-operative pain by record additional analgesics amount (rescue medication, mg) in PAR

SECONDARY OUTCOMES:
degree of post-operative nausea in post-anesthesia room (PAR) | 30 minutes
  Record the degree of nausea in PAR: mild, moderate, severe
degree of post-operative vomiting in post-anesthesia room (PAR) | 30 minutes
  Record the degree of vomiting in PAR: mild, moderate, severe
post-operative blood pressure in post-anesthesia room (PAR) | 0 minutes
  Record the blood pressure(mmHg) in PAR
post-operative systolic blood pressure in post-anesthesia room (PAR) | 0 minutes
  Record the systolic blood pressure(mmHg) in PAR
post-operative systolic blood pressure in post-anesthesia room (PAR) | 30 minutes
  Record the systolic blood pressure(mmHg) in PAR
post-operative diastolic blood pressure in post-anesthesia room (PAR) | 30 minutes
  Record the diastolic blood pressure(mmHg) in PAR
post-operative heart rate in post-anesthesia room (PAR) | 0 minutes
  Record the heart rate (beat/min) in PAR
post-operative heart rate in post-anesthesia room (PAR) | 30 minutes
  Record the heart rate (beat/min) in PAR
post-operative pulse oximeter in post-anesthesia room (PAR) | 0 minutes
  Record the pulse oximeter(SpO2; %) in PAR
postoperative pulse oximeter in post-anesthesia room (PAR) | 30 minutes
  Record the pulse oximeter(SpO2; %) in PAR
Numerical Rating Score (NRS) for pain score in ward | 1 hour after transferring to ward
  Record the degree of post-operative pain by Numerical Rating Scale (NRS)(0-10; 0= no pain; 10=pain as bad as can be)
Numerical Rating Score (NRS) for pain score in ward | 2 hours after transferring to ward
  Record the degree of post-operative pain by Numerical Rating Scale (NRS)(0-10; 0= no pain; 10=pain as bad as can be)
Numerical Rating Score (NRS) for pain score in ward | 4 hours after transferring to ward
  Record the degree of post-operative pain by Numerical Rating Scale (NRS)(0-10; 0= no pain; 10=pain as bad as can be)
Numerical Rating Score (NRS) for pain score in ward | 8 hours after transferring to ward
  Record the degree of post-operative pain by Numerical Rating Scale (NRS)(0-10; 0= no pain; 10=pain as bad as can be)
Numerical Rating Score (NRS) for pain score in ward | 24 hours after transferring to ward
  Record the degree of post-operative pain by Numerical Rating Scale (NRS)(0-10; 0= no pain; 10=pain as bad as can be)
total analgesics requirement in ward | 24hr after transferring to ward
  Record total analgesic requirement (mg) in ward

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-cherng Yu, MD, Study Chair — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Numerical rating scale, rescue analgesic amount